CLINICAL TRIAL: NCT02492854
Title: Standard Versus PICO Dressings in Lower-Extremity Bypass Patients
Acronym: PICO-LEB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided not to proceed with the major amendment and switching to the new generation of the device due to lack of funding.
Sponsor: Boston Medical Center (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-33618
Record Dates: First submitted 2015-06-24; First posted 2015-07-09 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Of Bypass Graft of the Extremities; Peripheral Arterial Disease; Vascular Diseases; Cardiovascular Diseases
Keywords: Lower Extremity Bypass; Surgical Site Infection; Wound Dressing; Negative Pressure Wound Dressing
MeSH Terms: conditions — Peripheral Arterial Disease; Vascular Diseases; Cardiovascular Diseases; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Sterile Gauze Dressings (Active Comparator): In this arm, pts. will be randomized to receive standard sterile gauze dressing post-operatively.
  Interventions: Other: Sterile Gauze Dressings
- PICO Negative Pressure Dressings (Experimental): In this arm, pts. will be randomized to receive PICO single-use negative pressure dressings.
  Interventions: Device: PICO Single-Use Negative Pressure Dressings

INTERVENTIONS:
Device: PICO Single-Use Negative Pressure Dressings — Negative pressure wound therapy (NPWT), over the past several years, has provided a way to post-operatively manage complex wounds. This is a therapy with potential to decrease rates of SSIs post-LE bypass. Unlike standard gauze dressings, negative pressure wound therapy provides a sealed, moist environment and shuttles fluid away from the wound. A suctioning unit applies even, negative pressure (typically -80 to -120 mmHg) and exudate is suctioned and collected in a control unit. The investigators would like to investigate the efficacy of PICO (Smith&Nephew), a single-use one-step wound dressing which is effective for 7 days. It is lightweight and uses a small hand-held vacuum pump, both of which allow for ease of use. PICO has been FDA-approved.
  Arms: PICO Negative Pressure Dressings
Other: Sterile Gauze Dressings — Current standard-of-care dressings used to cover surgical wounds post-operatively.
  Arms: Standard Sterile Gauze Dressings

SUMMARY:
The objective of this study is to compare the effectiveness of standard moist dressings and PICO single-use negative pressure dressings in post-operative lower extremity bypass patients. This study will compare the dressings' ability to decrease swelling, decrease post-operative infection, and improve mobility and quality of life measures.

Subjects will be asked to participate in this study because they will undergo a lower extremity bypass using the ipsilateral great saphenous vein. Subjects will then be randomized to two post-operative treatment groups. One group will receive standard sterile gauze and the other will receive PICO single-use negative pressure dressings. Both groups will be assessed for study measures in follow-up visits as clinically indicated up to 1 year with the 30 day timepoint as the primary outcome for study measures.

DETAILED DESCRIPTION:
Post-operative infection after lower extremity bypass operations (LEB) can lead to devastating consequences. A systematic review of lower-extremity (LE) re-vascularization cases using the American College of Surgeons National Surgical Quality Improvement Program (ACS-NSQIP) found that 11.1% of patients were diagnosed with surgical site infections (SSI). Another main issue in LEB is swelling, which occurs in about 70% of these patients and leads to increased pressure along the leading edges of often-long wounds.

A wide variety of methods to decrease these post-operative consequences are currently part of standard practice. These techniques include covering incision sites with sterile gauze dressing, elevating the leg, and wrapping with pressure dressings. Patients are then instructed to change dressings themselves at home. However, SSI rates demonstrate that these are only partially effective measures, and there remains room to improve post-operative management of infection and swelling.

Negative pressure wound therapy (NPWT), over the past several years, has provided a way to post-operatively manage complex wounds (see device description). PICO single-use negative pressure dressings have been examined in previous studies. However, these were either case series, for chronic wounds, or for non-vascular procedures. The effectiveness of PICO versus standard dressings in LEB has yet to be determined in a prospective, comparative study. Results will indicate whether PICO should be included standard post-operative care of lower-extremity bypass patients. This study is designed to compare PICO and standard care, and determine which offers the best outcomes of decreased days to ambulation and post-operative wound complications.

ELIGIBILITY:
Inclusion Criteria:

* Age > 35 years
* Patient to undergo lower extremity bypass using ipsilateral great saphenous vein harvest
* Willing to comply with protocol, attend follow-up appointments, complete all study assessments, and provide written informed consent.

Exclusion Criteria:

* Patients who received an investigational drug for peripheral arterial disease within 4 weeks of screening or who participated in another non-observational clinical trial in the prior 30 days
* Inability or refusal to provide informed consent
* Pregnancy or lactation
* Current immune-suppressive medication, chemotherapy, or radiation therapy
* Any infrainguinal revascularization procedure on index leg within 12 weeks prior to treatment
* Life expectancy of less than 2 years
* Prior leg bypass on the ipsilateral limb

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Siracuse, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PICO Negative Pressure Dressings: In this arm, pts. will be randomized to receive PICO single-use negative pressure dressings.
  PICO Single-Use Negative Pressure Dressings: Negative pressure wound therapy (NPWT), over the past several years, has provided a way to post-operatively manage complex wounds. This is a therapy with potential to decrease rates of surgical-site infections (SSIs) post-lower extremity (LE) bypass. Unlike standard gauze dressings, negative pressure wound therapy provides a sealed, moist environment and shuttles fluid away from the wound. A suctioning unit applies even, negative pressure (typically -80 to -120 mmHg) and exudate is suctioned and collected in a control unit. The investigators would like to investigate the efficacy of PICO (Smith&Nephew), a single-use one-step wound dressing which is effective for 7 days. It is lightweight and uses a small hand-held vacuum pump, both of which allow for ease of use. PICO has been FDA-approved.
Period: Overall Study
Arm/Group | Standard Sterile Gauze Dressings | PICO Negative Pressure Dressings
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Sterile Gauze Dressings | PICO Negative Pressure Dressings | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (8.3) | 60.3 (12.1) | 60.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Composite Score for Post-Operative Recovery
Description: The primary endpoint is lower-extremity bypass post-operative recovery that is free of major complications at 30 days post operation. This will be measured by a composite score based on three outcomes- leg swelling, ambulation, and infection (defined as antibiotics being prescribed). Each will be assigned a 0 if not present or a 1 if present and then summed for the composite score. The range can be from 0 to 3 with higher scores associated with more complications associated with surgical site infection.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Standard Sterile Gauze Dressings | PICO Negative Pressure Dressings
Number analyzed (Participants) | 5 | 3
scores on a scale | 0.80 (0.45) | 0.33 (0.58)

2. Secondary Outcome: Function and Quality of Life Based on the Vascular Quality of Life Survey
Description: The Vascular Quality of Life (VascuQol) survey is a 25 item instrument that is used to assess function and quality of life. Every item has a 7-point response scale ranging from 1 (worst) to 7 (best). The range of scores is 25 to 175. Higher scores are associated with higher function and quality of life.
Time Frame: 1 year
Population: For the Standard Sterile Gauze Dressing arm, data were not collected for 3 of the 5 participants as the study was terminated before 1 year of follow-up for those participants.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Standard Sterile Gauze Dressings | PICO Negative Pressure Dressings
Number analyzed (Participants) | 2 | 3
scores on a scale | 121.50 (7.78) | 144.67 (6.66)

3. Other Pre Specified Outcome: Resource Utilization in Dollars [Composite Measure]
Description: The resource utilization will be calculated from costs associated with the length of stay and discharge to rehabilitation centers which will be abstracted form the medical records.
Time Frame: 1 year
Population: Since the study was terminated, this outcome measure was not assessed for any of the participants.
Arm/Group | Standard Sterile Gauze Dressings | PICO Negative Pressure Dressings
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Standard Sterile Gauze Dressings | PICO Negative Pressure Dressings
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/5 | 1/3
Other Adverse Events (participants affected / at risk) | 3/5 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Sterile Gauze Dressings (N=5) | PICO Negative Pressure Dressings (N=3)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgical Site Infection (Infections and infestations) | 0 (0) | 1 (1)
Hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abcess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infected bypass graft (Infections and infestations) | 0 (0) | 1 (1)
Acute chest pain (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Sterile Gauze Dressings (N=5) | PICO Negative Pressure Dressings (N=3)
Cellulites (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peripheral arterial disease (Vascular disorders) | 1 (1) | 0 (0)
Altered mental status (Psychiatric disorders) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Serosanguisous discharge (Infections and infestations) | 0 (0) | 1 (1)
Redness and swellig (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The Covid pause halted participant enrollment and the PI decided not to proceed with the major amendment and switching to the new generation of the device due to lack of funding. This resulted in study termination, a small number of subjects for analysis, and incomplete data collection for the outcome measure designed to be collected at 1 year.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT02492854/Prot_SAP_000.pdf